CLINICAL TRIAL: NCT07341542
Title: Assessment of Surgical Margins in Breast Cancer Patients Using the Histolog Scanner: A Pilot Prospective Study in the Czech Republic
Brief Title: A Prospective Clinical Study Investigating the Use of the Histolog Scanner for Intraoperative Assessment of Surgical Margins in Patients Undergoing Breast-conserving Surgery for Histologically Confirmed Breast Cancer. The Histolog Scanner Operates on the Principle of Confocal Microscop
Status: Not yet recruiting | Type: Observational
Sponsor: Silesian Hospital in Opava (Other)
Responsible Party: Principal Investigator, Jan Žatecký, Jan Žatecký, MD, PhD, Silesian Hospital in Opava
Other Study IDs: EK SNO 435/2026
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; histolog scanner; surgical margins; breast-conserving surgery
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Histolog scanner — The aim of the project is a prospective pilot evaluation in a cohort of 20 patients to determine whether the use of the Histolog Scanner may, in the future, reduce the number of reoperations by identifying positive surgical margins already during the initial procedure.The specimen will subsequently be sent for standard histopathological assessment; therefore, the use of this method does not pose any risk to the patient, as the diagnostic and therapeutic pathway for breast cancer will not be altered.

SUMMARY:
A prospective clinical study investigating the use of the Histolog Scanner for intraoperative assessment of surgical margins in patients undergoing breast-conserving surgery for histologically confirmed breast cancer. The Histolog Scanner operates on the principle of confocal microscopy and enables non-destructive evaluation of specimen margins. The specimen will subsequently be sent for standard histopathological assessment; therefore, the use of this method does not pose any risk to the patient, as the diagnostic and therapeutic pathway for breast cancer will not be altered.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer confirmed by core-cut biopsy
* indication for breast-conserving surgery by a multidisciplinary team
* surgical therapy in Silesian Hospital in Opava during the study period

Exclusion Criteria:

* 0

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for breast-conserving surgery in Silesian Hospital in Opava for breast cancer confirmed by core-cut biopsy.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of reoperation rate (%) | 4 months
  Intraoperative assessment of the surgical specimen using the Histolog Scanner in breast cancer patients undergoing breast-conserving surgery reduces the likelihood of reoperation for an R1 resection, i.e., tumor involvement at the surgical margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Silesian Hospital in Opava, Opava, Czechia

IPD SHARING:
Plan to Share IPD: No